CLINICAL TRIAL: NCT05646316
Title: A Phase III Trial Of The Impact Of Sentinel Lymph Node Mapping On Patient Reported Lower Extremity Limb Dysfunction In Endometrial Cancer
Brief Title: Impact of Sentinel Lymph Node Mapping on Patient Reported Lower Extremity Limb Dysfunction in Stage I Endometrial Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NRG-CC010; NCI-2022-05090 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-CC010 (Other: NRG Oncology); NRG-CC010 (Other: DCP); NRG-CC010 (Other: CTEP); UG1CA189867 (NIH)
Record Dates: First submitted 2022-12-02; First posted 2022-12-12 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Stage I Uterine Corpus Carcinoma or Carcinosarcoma AJCC v8
MeSH Terms: conditions — Carcinosarcoma | interventions — Specimen Handling; X-Rays; Biopsy; Indocyanine Green; Minimally Invasive Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (sentinel lymph node mapping) (Experimental): Patients receive ICG dye via injection and undergo sentinel lymph node mapping and excision during standard minimally invasive hysterectomy. Lymph nodes around the uterus may be removed if the mapping and excision cannot be completed. Successful mapping requires no additional removal of lymph nodes. Patients also undergo imaging as clinically indicated and optional blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Diagnostic Imaging Testing; Procedure: Excisional Biopsy; Drug: Indocyanine Green Solution; Procedure: Minimally Invasive Surgery; Procedure: Pelvic Lymphadenectomy; Other: Questionnaire Administration; Procedure: Sentinel Lymph Node Mapping
- Arm 2 (sentinel lymph node mapping, pelvic lymphadenectomy) (Experimental): Patients receive ICG dye via injection and undergo sentinel lymph node mapping and excision during standard minimally invasive hysterectomy. Additional lymph nodes around the uterus are removed per standard of care. Patients also undergo imaging as clinically indicated and optional blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Diagnostic Imaging Testing; Procedure: Excisional Biopsy; Drug: Indocyanine Green Solution; Procedure: Minimally Invasive Surgery; Procedure: Pelvic Lymphadenectomy; Other: Questionnaire Administration; Procedure: Sentinel Lymph Node Mapping

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Diagnostic Imaging Testing — Undergo imaging
  Other Names: Diagnostic Imaging; Medical Imaging
Procedure: Excisional Biopsy — Undergo sentinel lymph node excision
  Other Names: Biopsy, Excisional; surgical biopsy
Drug: Indocyanine Green Solution — Given via injection
  Other Names: IC-GREEN; ICG Solution
Procedure: Minimally Invasive Surgery — Undergo minimally invasive hysterectomy
  Other Names: Minimally-Invasive Surgery; Surgery, Minimally Invasive
Procedure: Pelvic Lymphadenectomy — Undergo pelvic lymphadenectomy
  Other Names: Excision Pelvic Lymph Nodes; Pelvic Lymph Node Dissection
Other: Questionnaire Administration — Ancillary studies
Procedure: Sentinel Lymph Node Mapping — Undergo sentinel lymph node mapping
  Other Names: Sentinel Lymph Node Imaging

SUMMARY:
This phase III trial compares the effect of sentinel lymph node mapping to standard lymph node dissection in reducing the risk of swelling in the legs (lymphedema) in patients undergoing a hysterectomy for stage I endometrial cancer. Standard lymph node dissection removes lymph nodes around the uterus during a hysterectomy to look for spread of cancer from the uterus to nearby lymph nodes. Sentinel lymph node mapping uses a special dye and camera to look for cancer that may have spread to nearby lymph nodes. Comparing the results of the procedures may help doctors predict the risk of long-term swelling in the legs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the rates of lower extremity limb dysfunction (defined as a >= 4-point increase in Gynecologic Cancer Lymphedema Questionnaire [GCLQ] symptom score from baseline) in patients with apparent uterine confined endometrial cancer randomized to one of two lymphatic assessment strategies at time of hysterectomy:

Ia. Sentinel lymph node mapping and excision followed by side-specific lymphadenectomy on sides without a sentinel lymph node (SLN) identified according to a National Comprehensive Cancer Network (NCCN) guidelines approved algorithm (Arm 1); Ib. Sentinel lymph node mapping and excision according to an NCCN Guidelines approved algorithm followed by bilateral pelvic +/- para-aortic lymphadenectomy (Arm 2).

SECONDARY OBJECTIVE:

I. To compare changes in lower extremity limb circumference in patients with apparent uterine confined endometrial cancer randomized to one of two lymphatic assessment strategies at time of hysterectomy.

II. To validate the test characteristics of a SLN mapping algorithm including SLN detection rates, rate of perioperative complications, rate of identifying lymphatic metastases, and detection of micrometastases using pathologic ultra-staging.

EXPLORATORY OBJECTIVES:

I. To compare adjuvant therapy decisions in patients with apparent uterine confined endometrial cancer randomized to one of two lymphatic assessment strategies at time of hysterectomy.

II. To explore the impact of patient characteristics (age, body mass index [BMI], race), extent of lymph node dissection, and adjuvant therapy decisions (radiation, chemotherapy) on the development of lower extremity limb dysfunction - as well as their interaction with lymph node assessment strategies.

III. To evaluate the cost-effectiveness of SLN mapping with or without completion of lymphadenectomy for endometrial cancer.

SAFETY OBJECTIVE:

I. To compare progression free and overall survival in patients with apparent uterine confined endometrial cancer randomized to one of two lymphatic assessment strategies at time of hysterectomy.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1: Patients receive ICG dye via injection and undergo sentinel lymph node mapping and excision during standard minimally invasive hysterectomy. Lymph nodes around the uterus may be removed if the mapping and excision cannot be completed. Successful mapping requires no additional removal of lymph nodes.

ARM 2: Patients receive ICG dye via injection and undergo sentinel lymph node mapping and excision during standard minimally invasive hysterectomy. Additional lymph nodes around the uterus are removed per standard of care.

Patients in both arms also undergo imaging as clinically indicated and optional blood sample collection throughout the study.

After completion of study intervention, patients are followed every 3 months for one year and at 18 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of endometrial cancer based on endometrial sampling with a plan to undergo laparoscopic or robotic hysterectomy and lymphatic assessment as part of primary management. Biopsy must be performed within 90 days prior to registration
* Clinical stage I endometrial cancer based on the following diagnostic workup:

  * History/physical examination within 30 days prior to registration is reassuring for the absence of metastatic disease
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1 or 2
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry and, for patients treated in the United States (U.S.), authorization permitting release of personal health information
* Patients must speak English or Spanish

Exclusion Criteria:

* Patients whom the surgeon believes is not a candidate for pelvic lymphadenectomy due to medical comorbidities or other technical challenges (i.e. morbid obesity or prior surgery)
* History of chemotherapy or immunotherapy for the treatment of endometrial cancer. Progestin-containing therapies such as megestrol, medroxyprogesterone, or levonorgestrel-containing intrauterine device (IUD) are acceptable
* History of radiation to the pelvis, groin or lower extremities, or surgery to the pelvic lymph nodes or inguinal lymph nodes
* Patients who are going to undergo another elective surgery during the same operative event as their hysterectomy (i.e., sacrocolpopexy, cholecystectomy)
* Patients with severe, active co-morbidity defined as follows:

  * History of patient or provider identified lower extremity lymphedema
  * History of patient or provider identified chronic lower extremity swelling
  * History of lower extremity or pelvic deep venous thromboembolism within 90 days of registration
  * History of lower extremity cellulitis within 90 days of registration
  * For the bioimpedance sub study only: patients with implantable metal devices (i.e. defibrillator, metal joint replacements, etc.) will not be eligible to participate in the bioimpedance sub study but will be eligible to participate in the overall study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Estimated)
Dates: Start 2022-12-07 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of patient-reported lower extremity limb dysfunction | From 18 months post-hysterectomy after undergoing lymphatic assessment to 39 months
  The primary endpoint is the incidence of patient-reported lower extremity limb dysfunction at 18 months post-hysterectomy after undergoing lymphatic assessment according to a National Comprehensive Cancer Network guideline-based sentinel lymph node (SLN) mapping algorithm with or without completion of lymphadenectomy. The primary endpoint will be assessed using the Gynecologic Cancer Lymphedema Questionnaire (GCLQ) questionnaire. Surveys will be performed at enrollment (pre-surgery) and at 3, 6, 9, 12, and 18 months post-surgery. Patient-reported lower extremity limb dysfunction will be defined as an increase in GCLQ symptom score of at least four (4) points from baseline at any time during the 18 months follow-up. The primary null hypothesis will be evaluated with an intent-to-treat chi-squared test, adjusted for stratification factors. Proportional hazards modeling will be used to generate a hazard ratio and 95% confidence limits of Arm 1 versus Arm 2.

SECONDARY OUTCOMES:
The incidence of lymphedema by quantifiable lower extremity limb changes | From enrollment and at 3, 6, 9, 12, and 18 months after surgery
  Patients will undergo circumferential lower extremity limb measures at three locations along each leg. Change will be estimated as measurement at baseline subtracted from measurement at follow-up. This will be assessed in both legs separately.
The incidence of lymphedema by bioimpedance assessments (if available) | From enrollment and at 3, 6, 9, 12, and 18 months after surgery.
  Patients will undergo circumferential lower extremity limb measures at three locations along each leg. Change will be estimated as measurement at baseline subtracted from measurement at follow-up. This will be assessed in both legs separately. The SOZO device by ImpediMed provides an L-Dex score for each leg at each assessment point as each limb is at risk for lower extremity lymphedema.
Rate of successful bilateral SLN identification | At time of surgery
  Will be assessed in both, and only as the time of surgery.
Rate of successful identification of lymph node metastasis | At time of surgery
  Will be assessed in both, and only as the time of surgery. The rate of lymph node metastasis identification during surgery will be compared between groups, with either t-tests or chi-squared tests where appropriate.
Rate of perioperative complications | At time of surgery
  Will be assessed in both arms separately, and only as the time of surgery. The rate of perioperative complications during surgery will be compared between groups, with either t-tests or chi-squared tests where appropriate.

OTHER OUTCOMES:
Adjuvant therapy decisions | Up to 24 months
  Adjuvant therapy decisions will be compared for patients according to study arm allocation after accounting for tumor characteristics, stage, and patient demographics to determine whether lymph node mapping strategies was associated with a difference in adjuvant therapy choice.
Incremental cost-effectiveness ratio (ICER) of a SLN mapping algorithm | From enrollment and at 3, 6, 9, 12, and 18 months after surgery
  To determine the ICER of a SLN mapping algorithm with or without full lymphadenectomy for endometrial cancer using the European Quality of Life 5 Dimensions 3 Level Version, medical records (EQ-5D-5L), and questionnaire to gather resource utilization for lymphedema treatment. The visual analog scale and index scores from the EQ-5D-DL will be calculated at baseline and change scores corresponding at each collected follow-up time point then compared between treatment arms using a t-test with a 2-sided significance level of 0.05. At each time point, the EQ-5D-5L is obtained, and quality of life related utility scores will be calculated from the EQ-5D-5L. A mean utility score and confidence intervals will be used for cost-effective modeling. Quality-adjusted life years are calculated as the weighted sum of survival time and quality of life-based utilities. A Markov model will be used to model cost for this analysis.
Progression free survival | The duration of time from study entry to time of progression or death, whichever occurs first, or date of last contact if neither progression nor death has occurred, assessed at 2 years after enrollment
  This endpoint is not expected to be sufficiently powered for a definitive comparison and will therefore be treated as supportive evidence.
Overall survival | Duration of time from study entry to time of death or the date of last contact, assessed at 2 years after enrollment
  This endpoint is not expected to be sufficiently powered for a definitive comparison and will therefore be treated as supportive evidence.

CONTACTS AND LOCATIONS:
Overall Officials: Edward J Tanner, Principal Investigator — NRG Oncology
Locations (54):
- United States (54):
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - UM Sylvester Comprehensive Cancer Center at Doral, Doral, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Augusta University Medical Center, Augusta, Georgia
  - Northwestern University, Chicago, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - IU Health North Hospital, Carmel, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - West Jefferson Medical Center, Marrero, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - LSU Healthcare Network / Metairie Multi-Specialty Clinic, Metairie, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Mercy Hospital Springfield, Springfield, Missouri
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Intermountain Health West End Clinic, Billings, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Fred and Pamela Buffett Cancer Center - Kearney, Kearney, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - Methodist Willowbrook Hospital, Houston, Texas
  - Houston Methodist West Hospital, Houston, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - Houston Methodist The Woodlands Hospital, The Woodlands, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia